CLINICAL TRIAL: NCT02651220
Title: Clinical End Point Study of Generic Adapalene and Benzoyl Peroxide Gel Versus Epiduo® Forte Gel in Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 71491705
Record Dates: First submitted 2016-01-05; First posted 2016-01-08 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adapalene and Benzoyl Peroxide Gel, 0.3%/2.5% w/w (Experimental)
  Interventions: Drug: Adapalene and Benzoyl Peroxide Gel
- Epiduo® Forte Gel 0.3%/2.5% w/w (Active Comparator)
  Interventions: Drug: Epiduo® Forte Gel
- Placebo (vehicle) Topical Gel (Placebo Comparator)
  Interventions: Drug: placebo gel

INTERVENTIONS:
Drug: Epiduo® Forte Gel — Adapalene and Benzoyl Peroxide Gel, 0.3%/2.5% w/w
  Arms: Epiduo® Forte Gel 0.3%/2.5% w/w
Drug: Adapalene and Benzoyl Peroxide Gel — Adapalene and Benzoyl Peroxide Gel, 0.3%/2.5% w/w
  Arms: Adapalene and Benzoyl Peroxide Gel, 0.3%/2.5% w/w
Drug: placebo gel — vehicle used as placebo
  Arms: Placebo (vehicle) Topical Gel

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Multiple-Site Clinical Study to Evaluate the Therapeutic Equivalence and Safety of adapalene and benzoyl peroxide gel, 0.3%/2.5% (Actavis Laboratories UT, Inc.) to Epiduo® Forte (adapalene and benzoyl peroxide) gel 0.3%/2.5% (Galderma) in the treatment of Acne Vulgaris

DETAILED DESCRIPTION:
Up to 1000 patients 12 to 40 years of age inclusive will be enrolled to have 870 patients in the modified intent-to-treat (mITT) population and 579 patients in the per-protocol (PP) population. The primary inclusion criteria are the presence of ≥ 20 inflammatory lesions (papules and pustules) and ≥ 25 non-inflammatory lesions (opened and closed comedones) and ≤ 2 nodulocystic lesions (i.e., nodules and cysts) on the face and an Investigator's Global Assessment (IGA) score of 3 or 4.

Eligible patients will be randomized in a 1:1:1 ratio to one of the three treatments (Test, Reference or Placebo) on Visit 1. Patients will be instructed to apply the first treatment on the evening of enrollment into the study and then continue to apply once daily for the next 83 days (for a total 84 days). Patients will attend the following scheduled clinic visits:

* Visit 1 - Screening/Baseline: Day 1
* Visit 2 - Interim Visit: Day 28 ± 4
* Visit 3 - Interim Visit: Day 56 ± 4
* Visit 4 - End of Study: Day 85 ± 4 Efficacy evaluations will be based on dermatological assessments in the clinic. The primary statistical analyses of interest are (1) the percent change from baseline to Week 12 in the number of inflamed (papules/pustules) lesions and non-inflamed (open and closed comedones) lesions. In addition, patients will also be evaluated by the Investigator to determine "Clinical Success" or "Clinical Failure" at Week 12

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female, ≥ 12 and ≤ 40 years of age with a clinical diagnosis of acne vulgaris.
2. Signed informed consent form that meets all criteria of current FDA regulations. For a patient considered to be a minor in the state he/she lives and is enrolled, the patient parent or legal guardian will be required to sign the consent form and the patient will sign an IRB approved "assent to participate" form.
3. Females of child bearing potential must not be pregnant or lactating at Visit 1 (as confirmed by a negative urine pregnancy test with a sensitivity of less than 25 mlU/mL or equivalent units of human chorionic gonadotropin). Women of childbearing potential must agree to the use of a reliable method of contraception (e.g., total abstinence, IUD, a double-barrier method [such as condom plus diaphragm with spermicide], oral, transdermal, injected or implanted non- or hormonal contraceptive), throughout the study. If the female is using a hormonal contraceptive, the same product must be taken for 3 months prior to Visit 1 and must agree not to replace with some other hormonal contraceptives during the study. A sterile sexual partner is not considered an adequate form of birth control.

   All females will be considered to be of childbearing potential unless they:
   * Are post-menopausal, defined as women who have been amenorrheic for at least 12 consecutive months, without other known or suspected primary cause.
   * Have been sterilized surgically or who are otherwise proven sterile (i.e., total hysterectomy, or bilateral oophorectomy) with surgery at least 4 weeks prior to Screening. Tubal ligation will not be considered a surgically sterile method.

   Female patients of childbearing potential are defined as:
   * Females without prior hysterectomy, or who have had any evidence of menses in the past 12 months.
   * Females who have been amenorrhea for ≥ 12 months, but the amenorrhea is possibly due to other causes, including prior chemotherapy, anti-estrogens, or ovarian suppression.
4. Have facial acne vulgaris with: ≥ 20 inflammatory lesions (i.e., papules and pustules) and ≥ 25 non-inflammatory lesions (i.e., open and closed comedones) and ≤ 2 nodulocystic lesions (i.e., nodules and cysts).
5. Have an Investigator's Global Assessment (IGA) score of 3 or 4 (see Appendix A).
6. Willing to comply with the study requirements and restrictions including refraining from the use of all other topical acne medications or antibiotics during the 12 week treatment period.
7. Patients who use make-up must have used the same brands/types for a minimum period of 14 days before study entry and must agree to not change brand/type or frequency of use throughout the study.

Exclusion Criteria:

1. Patient has more than 2 facial nodular lesions; any nodules present will be documented but not included in the inflammatory and non-inflammatory lesion count for analysis.
2. Patient has active cystic acne.
3. Patient has acne conglobata, acne fulminans, or acne vulgaris requiring systemic treatment.
4. Patient has a skin condition that would interfere with the diagnosis or assessment of acne vulgaris (e.g., on the face: rosacea, dermatitis, psoriasis, squamous cell carcinoma, eczema, acneform eruptions caused by medications, steroid acne, steroid folliculitis, bacterial folliculitis).
5. Patients with excessive facial hair such as beards, sideburns, moustaches, etc. that would interfere with the diagnosis or assessment of acne.
6. Patients with tattoos or excessive facial scarring that, in the Investigator's opinion, may interfere with the evaluation of the patient's acne.
7. Patients with active facial sunburn, peeling from sunburn, or patients that will be exposed to excessive sunlight during the study.
8. Females who are pregnant, lactating or likely to become pregnant during the study.
9. History of allergy or hypersensitivity to adapalene, retinoids, benzoyl peroxide or history of any drug hypersensitivity or intolerance that, in the Investigator's opinion, would compromise the safety of the patient or the study.
10. Significant history or current evidence of chronic infectious disease, system disorder, organ disorder or other medical condition that, in the Investigator's opinion, would place the study participant at undue risk by participation.
11. Use of the following on the face within 1 month before Screening/Baseline:

    * Cryodestruction or chemodestruction
    * Dermabrasion
    * Photodynamic therapy
    * Acne surgery
    * Intralesional steroids
    * X-ray therapy
12. Use of the following within 1 month before Screening/Baseline:

    * Spironolactone
    * Systemic steroids
    * Systemic antibiotics
    * Systemic anti-inflammatory agents (the use of acetylsalicylic acid for prophylactic use up to 325 mg/day is allowed, provided that the patient is on a stable dose and the regimen will remain constant throughout the study). Acetaminophen will be allowed during the study with a maximum dose of 1g (i.e., 1000 mg) twice daily and for a maximum of 3 consecutive days (its use is not allowed within 1 week of each visit).
    * Systemic treatment for acne vulgaris (other than oral retinoids that require a 6 month washout), including anti-androgens.
13. Use of oral isotretinoin (Accutane®) or oral retinoids within 6 months, or therapeutic vitamin A supplements greater than 10,000 units/day (multivitamins are allowed).
14. Use of the following on the face within 2 weeks before Screening/Baseline:

    * Topical steroids
    * Topical retinoids
    * Topical zinc
    * Topical anti-inflammatory agents (including salicylic acid)
    * Topical antibiotics (including antibacterials)
    * Benzoyl peroxide
    * Any other topical over-the-counter preparations for acne treatment
15. Use of the following on the face within 1 week before Screening/Baseline:

    * Phototherapy devices for acne (e.g., ClearLightTM)
    * Medicated cleansers including adhesive cleansing strips
    * Cosmetic procedures (i.e., facials, peeling, comedone extraction) and alpha-hydroxy/glycolic acid
16. Receipt of any drug as part of a research study within 30 days.
17. Female patients taking hormonal contraceptives or oral estrogen for less than three months and those that plan to change the dosage regimen during the course of the study.
18. Previous participation in this study.
19. Employees of the Investigator or research center or their immediate family members.
20. Patients who are illiterate.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1001 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (18):
  - Site 103, Mesa, Arizona
  - Site 109, Tucson, Arizona
  - Site 112, Anaheim, California
  - Site 110, Long Beach, California
  - Site 111, Los Angeles, California
  - Site 104, San Diego, California
  - Site 113, West Covina, California
  - Site 101, Brandon, Florida
  - Site 119, Jacksonville, Florida
  - Site 114, Miami, Florida
  - Site 115, Miami, Florida
  - Site 116, Miramar, Florida
  - Site 102, Arlington Heights, Illinois
  - Site 105, Carmel, Indiana
  - Site 120, New Albany, Indiana
  - Site 107, Henderson, Nevada
  - Site 106, High Point, North Carolina
  - Site 108, Rhinelander, Wisconsin
- Belize (2):
  - Site 117, Belize City
  - Site 118, Belize City

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1001 patients were randomized, 24 did not receive any study medication.
Groups:
- Adapalene and Benzoyl Peroxide Gel, 0.3%/2.5% w/w: Generic: Adapalene and Benzoyl Peroxide Gel, 0.3%/2.5% w/w
- Epiduo® Forte Gel 0.3%/2.5% w/w: Reference: Epiduo® Forte Gel: Adapalene and Benzoyl Peroxide Gel, 0.3%/2.5% w/w
- Vehicle Topical Gel: Placebo gel: vehicle used as placebo
Period: Overall Study
Arm/Group | Adapalene and Benzoyl Peroxide Gel, 0.3%/2.5% w/w | Epiduo® Forte Gel 0.3%/2.5% w/w | Vehicle Topical Gel
Started | 337 | 335 | 329
Completed | 314 | 308 | 300
Not Completed | 23 | 27 | 29
Not completed — Adverse Event | 1 | 5 | 1
Not completed — Lost to Follow-up | 8 | 14 | 14
Not completed — Non-Compliance with Study Drug | 4 | 0 | 1
Not completed — Pregnancy | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 6 | 8
Not completed — Miscellaneous | 4 | 1 | 2
Not completed — Withdrawal by Parent/Guardian | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Data is presented here for the Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Adapalene and Benzoyl Peroxide Gel, 0.3%/2.5% w/w | Epiduo® Forte Gel 0.3%/2.5% w/w | Vehicle Topical Gel | Total
Number analyzed (Participants) | 332 | 323 | 322 | 977
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.5 (7.1) | 22.5 (7.1) | 22.5 (7.0) | 22.5 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 202 | 215 | 614
  Male | 135 | 121 | 107 | 363
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 139 | 148 | 134 | 421
  Not Hispanic or Latino | 193 | 175 | 188 | 556
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 0 | 3
  Asian | 25 | 18 | 16 | 59
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 111 | 114 | 123 | 348
  White | 186 | 187 | 175 | 548
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 3 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 12 in the Number of Inflamed Lesions.
Time Frame: 12 weeks
Population: Using the Per Protocol Population
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Adapalene and Benzoyl Peroxide Gel, 0.3%/2.5% w/w | Epiduo® Forte Gel 0.3%/2.5% w/w | Vehicle Topical Gel
Number analyzed (Participants) | 285 | 281 | 277
percentage of change from baseline | -74.2 (25.0) | -73.0 (27.8) | -30.6 (32.7)
Statistical Analysis 1: Comparison: Adapalene and Benzoyl Peroxide Gel, 0.3%/2.5% w/w vs Epiduo® Forte Gel 0.3%/2.5% w/w; Test type: Equivalence — Bioequivalence was based on 90% confidence interval within 80-125%; Bioavailability = 100.28, 90% CI 2-sided [96.78 to 103.91]

2. Primary Outcome: Percent Change From Baseline to Week 12 in the Number of Non-inflamed Lesions.
Time Frame: 12 weeks
Population: Using the Per Protocol Population
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Adapalene and Benzoyl Peroxide Gel, 0.3%/2.5% w/w | Epiduo® Forte Gel 0.3%/2.5% w/w | Vehicle Topical Gel
Number analyzed (Participants) | 285 | 281 | 277
percentage of change from baseline | -65.4 (25.7) | -64.5 (26.0) | -25.5 (30.1)
Statistical Analysis 1: Comparison: Adapalene and Benzoyl Peroxide Gel, 0.3%/2.5% w/w vs Epiduo® Forte Gel 0.3%/2.5% w/w; Test type: Equivalence — Bioequivalence is based on 90% confidence interval within 80-125%; Bioavailability = 99.73, 90% CI 2-sided [96.04 to 103.56]

3. Secondary Outcome: Percentage of Patients With a Clinical Response of "Clinical Success" Using the Investigator's Global Assessment (IGA) at Week 12
Description: The Investigator's Global Assessment had to show a score of 0 (clear) or 1 (almost clear) to be considered a "Clinical Success".
  0= Clear skin with no inflammatory or non inflammatory lesions.
  1. Almost clear, rare non-inflammatory lesions with no more than one small inflammatory lesion.
  2. Mild severity; greater than Grade 1; some non inflammatory lesions with no more than a few inflammatory lesions (papules/pustules only, no nodular lesions).
  3. Moderate severity; greater than Grade 2; up to many non inflammatory lesions and may have some inflammatory lesions, but no more than one small nodular lesion.
  4. Severe; greater than Grade 3, up to many non inflammatory lesions and may have some inflammatory lesions, but no more than a few nodular lesions.
  5. Very severe, greater than Grade 4
Time Frame: 12 weeks
Population: Using the Modified Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Adapalene and Benzoyl Peroxide Gel, 0.3%/2.5% w/w | Epiduo® Forte Gel 0.3%/2.5% w/w | Vehicle Topical Gel
Number analyzed (Participants) | 331 | 321 | 321
Participants | 112 | 106 | 15
Statistical Analysis 1: Comparison: Adapalene and Benzoyl Peroxide Gel, 0.3%/2.5% w/w vs Vehicle Topical Gel; Test type: Superiority; p < 0.0001, ANOVA

ADVERSE EVENTS:
Time Frame: Up to at least 3 months
Arm/Group | Adapalene and Benzoyl Peroxide Gel, 0.3%/2.5% w/w | Epiduo® Forte Gel 0.3%/2.5% w/w | Vehicle Topical Gel
All-Cause Mortality (participants affected / at risk) | 0/332 | 0/323 | 0/322
Serious Adverse Events (participants affected / at risk) | 0/332 | 0/323 | 2/322
Other Adverse Events (participants affected / at risk) | 27/332 | 41/323 | 26/322
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adapalene and Benzoyl Peroxide Gel, 0.3%/2.5% w/w (N=332) | Epiduo® Forte Gel 0.3%/2.5% w/w (N=323) | Vehicle Topical Gel (N=322)
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapalene and Benzoyl Peroxide Gel, 0.3%/2.5% w/w (N=332) | Epiduo® Forte Gel 0.3%/2.5% w/w (N=323) | Vehicle Topical Gel (N=322)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Application site dryness (General disorders) | 0 (0) | 5 (8) | 1 (1)
Application site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Application site hypersensitivity (General disorders) | 0 (0) | 1 (1) | 0 (0)
Application site irritation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Application site pain (General disorders) | 1 (1) | 5 (6) | 0 (0)
Application site pruritus (General disorders) | 0 (0) | 2 (3) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple allergies (Immune system disorders) | 1 (2) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Chlamydial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 10 (10) | 6 (6)
Nasopharyngitis (Infections and infestations) | 7 (7) | 8 (8) | 5 (5)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vaginitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Musckuloskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Heachache (Nervous system disorders) | 4 (4) | 2 (3) | 3 (4)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic fluid collection (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin tightness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.